CLINICAL TRIAL: NCT04850859
Title: Morphological and Morphometric Study on Human Glenoid Cavity and Acetabulum With Correlation to Their Functions
Brief Title: Study on Human Glenoid Cavity and Acetabulum
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mary Milad Alkesan, Demonstrator at Anatomy and Embryology Department, Faculty of medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-21-04-07
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Glenoid Cavity; Acetabulum
Keywords: glenoid cavity; acetabulum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group of scapulae bones: Human adult dry scapulae bones 40 of unknown sex and age will be collected.
  Interventions: Other: measure various dimensions of the glenoid
- group of hip bones: Human adult dry hip bones 40 of unknown gender and age will be collected
  Interventions: Other: measure various dimensions of the acetabulum

INTERVENTIONS:
Other: measure various dimensions of the glenoid — measurement of Superior-Inferior glenoid diameter ,Anterior-Posterior glenoid diameter and study shape of the glenoid cavity .
  Groups: group of scapulae bones
Other: measure various dimensions of the acetabulum — measurement of transverse diameter of the acetabulum ,vertical diameter of the acetabulum, depth of the acetabulum ,Width of acetabular notch and study shape of anterior acetabular ridge and ends of lunate surface .
  Groups: group of hip bones

SUMMARY:
1 - study morphological and morphometric features of the glenoid cavity in human scapulae bone and its function.

2- study morphological and morphometric features of the acetabulum in human hip bone and its function.

DETAILED DESCRIPTION:
study morphological features of the glenoid cavity and to measure various dimensions of the glenoid in dry human scapulae bone and correlation to its function.

The knowledge of normal anatomical features and variations of the shape and size of glenoid cavity are prerequisites for complete understanding of the mechanics of shoulder joint, this information has clinical application in shoulder arthroplasty, gleno-humeral instability and rotator cuff tear management.

study morphological features of the acetabulum and to measure various dimensions of the acetabulum in dry human hip bone and correlation to its function.

Knowledge of the dimensions of acetabulum are vital to understand the mechanics of hip joint, and will assist the prosthetists to construct the suitable prostheses

ELIGIBILITY:
Inclusion Criteria:

* The scapulae with clear and intact glenoid cavity will be used for the study. The hip bones with clear and intact acetabulum will be used for the study

Exclusion Criteria:

* Bones with gross damage or anomalies will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: scapulae bones and hip bones will be collected at anatomy department of Sohag faculty of medicine
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
study morphological features of the glenoid cavity and measure various dimensions of the glenoid in dry human scapulae bone. | 2months following the start point of the study
  measurement of Superior-Inferior glenoid diameter ,Anterior-Posterior glenoid diameter by using Vernier caliper in millimeter with accuracy of 0.01mm
study morphological features of the acetabulum and measure various dimensions of the acetabulum in dry human hip bone. | 2months following the start point of the study
  measurement of transverse diameter of the acetabulum ,vertical diameter of the acetabulum, depth of the acetabulum ,Width of acetabular notch by using Vernier caliper in millimeter with accuracy of 0.01mm

CONTACTS AND LOCATIONS:
Overall Officials: Mary Milad Alkesan, Principal Investigator — Sohag University
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
because data will be collected from bones of unknown sex and age